CLINICAL TRIAL: NCT01246557
Title: Open Label Multi-center Pilot Phase I/II Non-controlled Clinical Trial to Assess Safety and Efficieecy of the Lenalidomide and Dexamethasone Association in Patients With Chronic Relapse or Treatment Resistant Lymphatic Leukemia Following Treatment Containing Fludarabine.
Brief Title: Study Assessing Safety and Efficiency of the Lenalidomide and Dexamethasone Combination in Patients With Chronic Lymphatic Leukemia (CLL) Relapsing or Resistant to Treatment
Acronym: LENDEX-LLC-09
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Hospital Universitari Vall d'Hebron Research Institute., Investigator
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENDEX-LLC-09; 2009-012571-95 (EudraCT Number)
Record Dates: First submitted 2010-09-30; First posted 2010-11-23 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Lymphatic Leukemia
Keywords: Patients with Chronic Lymphatic Leukemia relapsing or resistant to treatment
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide - Revlimid®: an analogue of thalidomide, is an immunomodulator agent with anti-angiogenic properties. The chemical name is 3-(4 ́-aminoisoindoline-1 ́ona)-1- piperidine-2,6-dione.
  REVLIMID® (lenalidomide) is available in capsules of 5 mg, 10 mg and 15 mg p.o.. Each capsule contains lenalidomide as active ingredient and the following non active ingredients: anhydrous lactose, microcrystalline cellulose, sodium croscarmellose and magnesium stearate.
  Other Names: REVLIMID®
Drug: Dexamethasone — Dexamethasone will be administered as 20 mg/day (on days 1 to 4) for oral administration.
  Other Names: Commercial drug according to standard clinical practices of the center.

SUMMARY:
Despite certain notable progress, treatment of patients with Chronic Lymphatic Leukemia (CLL) is still disappointing. Although thanks to the use of treatment of (immune) chemotherapy, mainly based on fludarabine, rituximab and alemtuzumab, the rate of complete response (CR) has increased from minus 10% observed when clorambucil was the core of the therapy to a 60-70%, with time all patients relapse and most of them die at the end due to the disease or to involvements related to the treatment. Progress when understanding the CLL biology have cleared a series of aspects: 1) there is a significant proportion of CLL cells actively copying themselves, contrary to the opinion that most of CLL cells are in G0 phase of the cell cycle; 2) Immune regulatory mechanism basically measured by T cells and NK cells have an important role in the continuous accumulation of CLL cells in the body; 3) Cells of the stroma are essential to maintain survival of CLL cells through a series of cytokines or chemokines. Under the light of this evidence, it is worth studying new treatment modes directed not only to CLL cells but also to the microenvironment and immune functions.

Lenalidomide is being investigated as treatment for several oncologic indications including myelodysplastic syndromes, multiple myeloma and non-Hodgkin lymphoma. Within the scope of CLL, it has been proved that lenalidomide is active in patients with relapsing / treatment resistant CLL patients. Forty five patients with relapsing CLL, 51% resistant to fludarabine, where included in a phase II study and were treated orally with 25 mg of lenalidomide on days 1 to 21 of a cycle of 28 days. The total response rate was of 47% with up to a 9% of complete responses.

The combination of lenalidomide with dexamethasone is being investigated in multiple myeloma and has revealed as a highly efficient treatment in relapsing/ treatment resistant patients as well as in those newly diagnosed. Bearing in mind that both drugs, lenalidomide and dexamethasone, are clinically active in CLL the investigators have designed a study with this combination in relapsing or treatment resistant patients following treatments containing fludarabine which do not meet the requirements for an intensive rescue treatment.

Given initial doses of 10 and 25 mg of lenalidomide daily may be associated with tumor lysis cases, it is proposed a low initial dose of lenalidomide in the first cycle 2.5mg., with further increases to prevent the occurrence of tumor lysis syndrome

ELIGIBILITY:
Inclusion Criteria:

The patients will have to meet the following inclusion criteria in order to be included in the study:

1. To understand and voluntarily sign an informed consent form.
2. To be ≥ 18 years old upon the signature of the informed consent form.
3. To be able to fulfill the visits program of the study and other protocol requirements.
4. To have a CLL documented diagnose (NCI/WG criteria) relapsing or resistant to at least one prior treatment and not to meet the requirements for an intensive rescue therapy. Prior treatment(s) will have to include fludarabine.
5. All prior anti-cancer therapies, including radiation, hormonal therapy and surgery, will have to be interrupted at leas 4 weeks before the treatment in this study.
6. Functional state 0-2 (ECOG).
7. Women with childbearing potential (FCBP) will have to:

   understand the teratogenic risk of the study drug. accept the simultaneous use of two reliable contraception methods or to practice the abstinence of heterosexual relations during the following periods of time related to this study: 1) during at least 4 weeks before starting the drug of the study; 2) while participating in the study; y 3) during at least 4 weeks following the interruption of the study. The two reliable contraceptive methods will have to include one highly effective (this is, intrauterine device (IUD), hormonal (pills injections or implants), tubal ligation, vasectomy of the partner) and an barrier effective additional method (this is, latex preservative, diaphragm, cervical cap). Women with a childbearing potential will have to visit a specialist in contraceptive methods if necessary.

   Before starting the drug under study: • Women with childbearing potential will have to undergo two negative pregnancy tests (sensibility of at least 25 mUI/ml) before starting the drug under study. The first test will take place at the visit date or within a period of 3 days before starting the drug under study and the second.The patient will not receive the drug until the investigator has verified that the results of the tests are negative.

   Men:
   * They will have to accept the use of latex preservatives during sexual relations with women with childbearing potential while they participate in the study and during at least one week following the interruption of the study, if it is women with childbearing potential (FCBP) and no use contraception.
   * They will have to accept to refrain from donating blood or semen during their participation in the study and during at least 28 days following the interruption of the study.
8. In the event of pregnancy or positive pregnancy test in a participant in the study, or the partner of a male participant in the study, during his participation, the drug under study will be immediately interrupted.
9. Capable of receiving Acetyl Salicylic Acid (100 or 300 mg) on a daily basis as prophylactic anticoagulation. (Patients who do not tolerate ASA may use acenocumarol or low molecular weight heparin).

Exclusion Criteria:

Patients will not have to fulfill any of the following exclusion criteria to be included in the study.

1. Any serious medical disorder, laboratory abnormality or psychiatric disease hindering the signature of the informed consent by the patient.
2. Pregnant women or in lactation period.
3. Any disorder, including the presence of laboratory abnormalities, which puts the patient at unacceptable risk if he/she participates in the study or hindered the capacity to understand the information of the study.
4. Use of any other experimental drug or therapy in the period of 28 days from the base visit.
5. Known hyper-sensibility to thalidomide.
6. Development of erythema nodosum if it is characterized by a descamative eruption while taken thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. A concurrent use of other agents or anticancer treatments.
9. HIV-positive or infectious hepatitis type A, B or C.
10. Candidates eligible for intensive rescue therapies (ex. R-CHOP plus alemtuzumab, allogenic transplant)
11. Richter transformation (active) or CNS participation (active)
12. Any of the following laboratory abnormalities:

    Neutrophil absolute count < 0.5 x 109/L Platelet count < 25 x 109/L Calculated Creatinine Clearance <50 mL/min Total serum bilirubin > higher normal limit (HNL) AST and ALT >3 x higher normal limit (HNL) Autoimmune non controlled hemolytic anemia or thrombocytopenia.
13. History of another neoplastic disease during ≥ 5 years unless base cells or epidermoid carcinoma in situ of cervix or breast recently treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the association of lenalidomide and dexamethasone in patients with relapsed or refractory CLL | At the finalization of the second cycle of the treatment of the last patient (average 5 months of last patient inclusion date)
  The first step will be an interim analysis of toxicity to determine the safety of the first lenalidomide cohort dosage (2.5 mg/day). This analysis will be performed after six subjects complete 3 months of treatment. A second analysis of toxicity will be performed after the second lenalidomide dosage cohort (six patients with 5mg/day) complete 3 months of treatment.

SECONDARY OUTCOMES:
To assess the efficacy of lenalidomide and dexamethasone in patients with Chronic Lymphocytic Leukemia (CLL) relapsing of resistant to treatment. | Average of 20 months from the last patient inclusion.
  Efficacy endpoint: Duration of response.
To assess the efficacy of lenalidomide and dexamethasone in patients with Chronic Lymphocytic Leukemia (CLL) relapsing of resistant to treatment. | Average of 9 months from the last patient inclusion.
  Efficacy endpoint: Time to response.
To assess the efficacy of lenalidomide and dexamethasone in patients with Chronic Lymphocytic Leukemia (CLL) relapsing of resistant to treatment. | Average of 20 months from the last patient inclusion.
  Efficacy endpoint: Progresion-free survival.
To assess the efficacy of lenalidomide and dexamethasone in patients with Chronic Lymphocytic Leukemia (CLL) relapsing of resistant to treatment. | Average of 20 months from the last patient inclusion.
  Efficacy endpoint: Treatment response.
To assess the efficacy of lenalidomide and dexamethasone in patients with Chronic Lymphocytic Leukemia (CLL) relapsing of resistant to treatment. | Average of 20 months from the last patient inclusion.
  Efficacy endpoint: Overall survival.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Centro Médico Teknon, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Valle Hebron, Barcelona, Barcelona
  - Hospital Clinico Universitario de Barcelona, Barcelona, Barcelona
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia